CLINICAL TRIAL: NCT05202938
Title: Energy MEtabolism of Septic Heart.
Brief Title: eMESH Struct. 2022-23
Acronym: eMESH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: eMESH struct. 2022-23; 2021-4012 (Other: CHUS ethical committee)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Septic Shock; Chronic Heart Failure
Keywords: Septic shock; Heart dysfunction; Positron emission tomography; Energy substrates (glucose, fatty acid, acetate); Mitochondrial activity
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 ml of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Septic shock with SIMD: SIMD+: 8 patients in septic shock (Sepsis-3-) with SIMD: ejection fraction (LVEF) < 45% in the first 48 hours of admission into the intensive care unit. No prior cardiac ultrasound or normal cardiac ultrasound values less than 2 years ago , or an ino-vasotropic infusion (milrinone, dobutamine, norepinephrine or epinephrine) required to obtain a LVEF ≥ 45%, or a drop of ≥ 20% compared to the LVEF value record ed less than 2 years ago.
  Interventions: Diagnostic Test: ultrasound cardiography; Diagnostic Test: FDG PET scan; Diagnostic Test: Palmitate PET scan; Diagnostic Test: Acetate PET scan; Diagnostic Test: Blood sampling
- Septic shock without SIMD: SIMD-: 8 patients in septic shock (Sepsis-3) without SIMD. Ejection fraction (LVEF) ≥ 45% with or without ino-vasotropic infusion (milrinone, dobutamine, norepinephrine or epinephrine), or similar to the LVEF recorded less than 2 years ago.
  Interventions: Diagnostic Test: ultrasound cardiography; Diagnostic Test: FDG PET scan; Diagnostic Test: Palmitate PET scan; Diagnostic Test: Acetate PET scan; Diagnostic Test: Blood sampling
- Acute Heart Failure with reduced Ejection Fraction: HFrEF: 8 patients with acutely reduced ejection fraction (LVEF) < 50%. with or without ino-vasotropic infusion (milrinone, dobutamine, norepinephrine or epinephrine) No prior cardiac ultrasound, or normal cardiac ultrasound values less than 2 years ago, or a drop of ≥ 20% compared to the LVEF recorded less than 2 years ago. No evidence of sepsis or septic shock.
  Interventions: Diagnostic Test: ultrasound cardiography; Diagnostic Test: FDG PET scan; Diagnostic Test: Palmitate PET scan; Diagnostic Test: Acetate PET scan; Diagnostic Test: Blood sampling
- Acute Heart Failure with preserved Ejection Fraction: HFpEF: 8 patients with acute heart failure and a preserved ejection fraction (ejection fraction (LVEF ≥ 50% or similar to normal cardiac ultrasound values recorded less than 2 years ago). No evidence of septic shock.
  Interventions: Diagnostic Test: ultrasound cardiography; Diagnostic Test: FDG PET scan; Diagnostic Test: Palmitate PET scan; Diagnostic Test: Acetate PET scan; Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: ultrasound cardiography — Ultrasound to check heart functions and systolic ejection fraction.
Diagnostic Test: FDG PET scan — FDG venous injection and positron emission tomography scan.
  Other Names: FDG positron emission tomography
Diagnostic Test: Palmitate PET scan — C11-Palmitate venous injection and positron emission tomography scan.
  Other Names: Palmitate positron emission tomography
Diagnostic Test: Acetate PET scan — C11-Acetate venous injection and positron emission tomography scan.
  Other Names: Acetate positron emission tomography
Diagnostic Test: Blood sampling — Collecting 20ml of venous blood.
  Other Names: Collecting blood sample

SUMMARY:
A flexible energy metabolism matched with the contractile needs of the muscle is essential to a normal heart. Loss of metabolic flexibility and cardiac systolic efficiency coexist in Sepsis-induced Myocardial Dysfunction (SIMD), a phenomenon attributed to mitochondrial dysfunction and mishandling of energy substrates. Cardiac positron emission tomography (PET) could allow to quantify non invasively the selection of energy substrates by the hearts in sepsis and will be associated in parallel with functional status (ultrasound cardiography), injury biomarkers, apelinergic and metabolomic blood profiles. Comparisons will be performed between septic and acute on chronic heart failures, with or without systolic dysfunction.

DETAILED DESCRIPTION:
Septic shock is both highly prevalent and morbid in the intensive care units. The mortality rate rises from 10-30% to 70-80% with sepsis-induced myocardial dysfunction (SIMD) occurence. SIMD is related to stress-induced cardiomyopathies and features bio-mechanistic components distinctive from chronic heart failure (CHF) traditionally attributed to a coronary disease. Dobutamine, a beta-adrenergic receptor agonist, is the inotrope drug actually recommended when cardiac index is too low, often in association with a mix of alpha-beta-adrenergic agonists like norepinephrine. In this context, dobutamine is marginally effective (1/3 responders), has potential deleterious impacts on function and viability of cardiomyocytes, and induces increased needs in cardiac energy metabolism. The healthy heart works almost exclusively on aerobic metabolism. While glucose is the essential fuel for brain and skeletal muscles, fatty acids through lipid oxidation are the main substrates for a normal resting heart (Randle cycle). This lipid oxidation is producing at least 70% of cardiac ATP, the balance is coming from glucose, with a marginal contribution from ketone bodies and lactate. The mitochondria is a cellular factory which produces more than 95% of body ATP. Mitochondria represent 30-40% of the cardiomyocyte total volume and consume oxygen to generate huge quantities of ATP/day by oxidative phosphorylation through 3 connective pathways: cytoplasmic glycolysis, Krebs cycle, and the mitochondrial electron transport chain inside the respiratory enzymes complex. Although a direct close relationship between myocardial metabolism homeostasis and function is not clearly established in normal condition, a compensatory equilibrium between fatty acid and glucose mitochondrial oxidations is a generally accepted concept. Indeed, the heart is omnivorous and can modulate fuel-substrates captation/utilization according to the physiological events (exercise, fast).That reprogramming capacity towards other various circumstances or pathological conditions is not guaranteed, with potential loss of metabolic flexibility. SIMD is highly prevalent in septic shock and is frequently indicative of a worsened outcome with increased mortality. Left ventricular systolic and diastolic dysfunctions are observed in 50% of acute sepsis within the first 48 hours after patient's admission. Animal experimental models can simulate human sepsis and SIMD by injecting endotoxin (LPS model) or feces in the abdominal cavity (cecal ligation puncture model), and with inflammatory cytokines, oxidative stress, nitric oxide and neutrophils as potential aggressors. Ventriculo-arterial and excitation-contraction decoupling are the hallmark of the contractile inefficiency observed in SIMD. Ca2+ handling (an ion molecule essential for heart function) in aberrant during sepsis and associated with impaired activation/phosphorylation and proteolytic cleavage increased of key regulators like heart troponin I. Resulting common cyto-histopathological damages are: myocardial apoptosis with focal necrosis, cardiac muscle edema, congestion, multiples inflammatory infiltrates, and mitochondrial structural insults with intra-myocardial accumulation of glycogen & lipids. The lathers could be a spillover effect of the cardiac metabolic shut-down consecutive to mitochondrial dysfunction. A decrease in fatty acid captation/oxidation has been documented in traditional CHF, not always offset by an enhanced use of glucose, but sometimes by an increased use of ketone bodies and lactates, and through an elevated myocardial proteolysis. This observation doesn't necessarily apply to sepsis and SIMD where cardiac energy metabolism is still a mystery. Systemic metabolic alterations in sepsis are complexe, with glycogenolysis and gluconeogenesis activations, insulinoresistance, and an increased lipolysis with enhanced fatty acid blood levels. In these conditions and in the heart, a drop of fatty acid oxidation is not necessarily compensated by an increased glucose use. Different denominations have been used to figure out these SIMD-induced metabolism disorders, the best being "metabolic-bioenergetic shut-down and stunning". In fact, sepsis induces a metabolic hurricane in bloodstream, vital organs and mitochondria, resulting in a significant rise of the rest energy expenditure. Dhainaut et al were first to demonstrate in 1987 a shift in the selection of energy fuels by myocardial tissues in septic shock patients. Both fatty acid and glucose uses were diminished by 4 and 2 times, respectively. However, this study addressed to suboptimally fluid resuscitated patients, who were in early acute hyperdynamic shock (< 6 hours). In experimental mouse models challenged with LPS or cecal ligation puncture, and adequate fluid resuscitation, the cardiac microperfusion is altered (i.e. malperfusion), and mitochondrial oxidative metabolism diminished, with an increase of glucose myocardial uptake. The apelin system is a family of endogenous peptides hormones (the apelins), not related to catecholamines, but with strong cardiovascular properties. This functional impact correlates with the constitutive expression of apelins and their receptor APJ in heart and vessels. Cardiac effects of apelins are characterized by an enhanced contractile force (systolic function), without chronotropic but with a lusitropic effect and a dromo-modulation. Another one impact of the apelins is on the cardiac utilization of metabolic energy substrates.

Apelins are facilitators-influencers glucose and fatty acid usage through recruitment of major specific carriers such as GLUT4 and FAT/CD36.

Research investigations: Which energy source is privileged by cardiac mitochondria in acute septic shock with or without myocardial dysfunction vs non-septic CHF ? Is this tentative shift/move of energy substrate's use related to muscle dysfunction or only reactive to the systemic environment ? and is it specific of sepsis or common to any non-specific myocardial damage ? Is this shift related to a particular biophenotype of the apelinergic system which is involved in the cardiovascular homeostasis ? and/or a distinctive alteration of the cardiac injury biomarkers ? Is the systemic environmental metabolomic affected toward a trending way during acute septic shock ?

Hypotheses: A myocardial positron emission tomography (PET) could allow to visualize and quantify non invasively energy supply selection of hearts in acute shock conditions related or not related to sepsis. Relationships can be found between PET profiles, sources of acute shock (sepsis vs non sepsis), functional data (ultrasound cardiography), cardiac injury specific biomarkers, apelinergic and metabolomic blood profiles.

Objectives: 1) To show the analytical value of the cardiac captation kinetic of 3 energy tracers (palmitate for fatty acids, FDG for glucose and acetate fpr mitochondrial activity), 2) To correlate PET data with myocardial (dys)function observed by US cardiography, 3) To evaluate the patients blood metabolomic profile in terms of products accumulation derived from a failure of energy substrates oxidation, 4) To measure and compare myocardial injury/ remodelling biomarkers (troponins, NT-proBNP, galectin-3) and the systemic endogenous apelin biophenotype.

Methods: 1) Prospective evaluative study of 4 groups of 8 patients in septic shock or in acute heart failure under hemodynamic support: i) a group with evidences of SIMD (US cardiography at the ICU ward in the first 48hrs: systolic ejection fraction < 45%), ii) a group in septic shock without evidence of SIMD, iii) a group with non-septic heart failure (systolic ejection fraction < 45% or cardiac insufficiency with reduced ejection fraction, iv) a group with non-septic (systolic ejection fraction < 50% or cardiac insufficiency with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in intensive care unit and coronary unit of the Sherbrooke hospital/CHUS.
* Accepts healthy volunteers: 4 to 6 age- and sex-matched HV will be recruited and imaged at the end of the inclusion window for the assessment of cardiac energy tracer's uptake and as ref. controls.

Exclusion Criteria:

* Pediatric patients
* Albumin allergy
* Moribund patients
* Patients too much unstable for the imaging procedure (clinical judgment)
* Unavailable tracers, staff, PET scan in a maximum delay of 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care unit and coronary unit of the Sherbrooke hospital/CHUS.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
FDG PET scan | 25 minutes
  Positron emission tomography with FDG radiotracer. It will report the glucose uptake by the heart.
Palmitate PET scan | 15 minutes
  Positron emission tomography with C11-palmitate radiotracer. It will report the fatty acid uptake by the heart.
Acetate PET scan | 10 minutes
  Positron emission tomography with C11-acetate radiotracer. It will report the acetate uptake by the heart.
Quantitative study of blood FDG:palmitate balance. | 20 minutes
  Measure of the blood FDG:palmitate balance by spectroscopy LC-MS and NMR.

SECONDARY OUTCOMES:
Measure of myocardial injury biomarkers. | 45 minutes
  Measure of blood myocardial injury biomarkers by immuno-enzymatic methods (Troponin T, NT-pro BNP, Galectin 3
Measure of apelinergics. | 45 minutes
  Measure of blood apelinergics (apelin-13 ,apelin-17, apelin-36 and ELABELA) by immuno-enzymatic methods.
Profiling of the systemic metabolomic. | 45 minutes
  Profiling of the systemic (blood) metabolomic by LC-MS and NMR. It will report metabolites in blood such as acetate, acetoacetate, acetone, 3-OH-butyrate, citrate, glutamate, lactate and pyruvate.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesur, MD PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Parrillo JE, Parker MM, Natanson C, Suffredini AF, Danner RL, Cunnion RE, Ognibene FP. Septic shock in humans. Advances in the understanding of pathogenesis, cardiovascular dysfunction, and therapy. Ann Intern Med. 1990 Aug 1;113(3):227-42. doi: 10.7326/0003-4819-113-3-227. PMID 2197912
- [Background] Merx MW, Weber C. Sepsis and the heart. Circulation. 2007 Aug 14;116(7):793-802. doi: 10.1161/CIRCULATIONAHA.106.678359. PMID 17698745
- [Background] Walley KR. Sepsis-induced myocardial dysfunction. Curr Opin Crit Care. 2018 Aug;24(4):292-299. doi: 10.1097/MCC.0000000000000507. PMID 29846206
- [Background] Taegtmeyer H, Young ME, Lopaschuk GD, Abel ED, Brunengraber H, Darley-Usmar V, Des Rosiers C, Gerszten R, Glatz JF, Griffin JL, Gropler RJ, Holzhuetter HG, Kizer JR, Lewandowski ED, Malloy CR, Neubauer S, Peterson LR, Portman MA, Recchia FA, Van Eyk JE, Wang TJ; American Heart Association Council on Basic Cardiovascular Sciences. Assessing Cardiac Metabolism: A Scientific Statement From the American Heart Association. Circ Res. 2016 May 13;118(10):1659-701. doi: 10.1161/RES.0000000000000097. Epub 2016 Mar 24. PMID 27012580
- [Background] Neely JR, Rovetto MJ, Oram JF. Myocardial utilization of carbohydrate and lipids. Prog Cardiovasc Dis. 1972 Nov-Dec;15(3):289-329. doi: 10.1016/0033-0620(72)90029-1. No abstract available. PMID 4564017
- [Background] Krishnagopalan S, Kumar A, Parrillo JE, Kumar A. Myocardial dysfunction in the patient with sepsis. Curr Opin Crit Care. 2002 Oct;8(5):376-88. doi: 10.1097/00075198-200210000-00003. PMID 12357104
- [Background] Antonucci E, Fiaccadori E, Donadello K, Taccone FS, Franchi F, Scolletta S. Myocardial depression in sepsis: from pathogenesis to clinical manifestations and treatment. J Crit Care. 2014 Aug;29(4):500-11. doi: 10.1016/j.jcrc.2014.03.028. Epub 2014 Apr 5. PMID 24794044
- [Background] Rudiger A, Singer M. Mechanisms of sepsis-induced cardiac dysfunction. Crit Care Med. 2007 Jun;35(6):1599-608. doi: 10.1097/01.CCM.0000266683.64081.02. PMID 17452940
- [Background] Lopaschuk GD. Metabolic Modulators in Heart Disease: Past, Present, and Future. Can J Cardiol. 2017 Jul;33(7):838-849. doi: 10.1016/j.cjca.2016.12.013. Epub 2016 Dec 21. PMID 28279520
- [Background] Karwi QG, Uddin GM, Ho KL, Lopaschuk GD. Loss of Metabolic Flexibility in the Failing Heart. Front Cardiovasc Med. 2018 Jun 6;5:68. doi: 10.3389/fcvm.2018.00068. eCollection 2018. PMID 29928647
- [Background] Pascual F, Coleman RA. Fuel availability and fate in cardiac metabolism: A tale of two substrates. Biochim Biophys Acta. 2016 Oct;1861(10):1425-33. doi: 10.1016/j.bbalip.2016.03.014. Epub 2016 Mar 16. PMID 26993579
- [Background] Doenst T, Nguyen TD, Abel ED. Cardiac metabolism in heart failure: implications beyond ATP production. Circ Res. 2013 Aug 30;113(6):709-24. doi: 10.1161/CIRCRESAHA.113.300376. PMID 23989714
- [Background] Drosatos K, Lymperopoulos A, Kennel PJ, Pollak N, Schulze PC, Goldberg IJ. Pathophysiology of sepsis-related cardiac dysfunction: driven by inflammation, energy mismanagement, or both? Curr Heart Fail Rep. 2015 Apr;12(2):130-40. doi: 10.1007/s11897-014-0247-z. PMID 25475180
- [Background] Carre JE, Singer M. Cellular energetic metabolism in sepsis: the need for a systems approach. Biochim Biophys Acta. 2008 Jul-Aug;1777(7-8):763-71. doi: 10.1016/j.bbabio.2008.04.024. Epub 2008 Apr 23. PMID 18482575
- [Background] Mangmool S, Denkaew T, Parichatikanond W, Kurose H. beta-Adrenergic Receptor and Insulin Resistance in the Heart. Biomol Ther (Seoul). 2017 Jan 1;25(1):44-56. doi: 10.4062/biomolther.2016.128. PMID 28035081
- [Background] Ehrman RR, Sullivan AN, Favot MJ, Sherwin RL, Reynolds CA, Abidov A, Levy PD. Pathophysiology, echocardiographic evaluation, biomarker findings, and prognostic implications of septic cardiomyopathy: a review of the literature. Crit Care. 2018 May 4;22(1):112. doi: 10.1186/s13054-018-2043-8. PMID 29724231
- [Background] Bertrand C, Valet P, Castan-Laurell I. Apelin and energy metabolism. Front Physiol. 2015 Apr 10;6:115. doi: 10.3389/fphys.2015.00115. eCollection 2015. PMID 25914650
- [Background] Reddy YN, Borlaug BA. Heart Failure With Preserved Ejection Fraction. Curr Probl Cardiol. 2016 Apr;41(4):145-88. doi: 10.1016/j.cpcardiol.2015.12.002. Epub 2015 Dec 9. PMID 26952248
- [Result] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Result] Parker MM, Shelhamer JH, Bacharach SL, Green MV, Natanson C, Frederick TM, Damske BA, Parrillo JE. Profound but reversible myocardial depression in patients with septic shock. Ann Intern Med. 1984 Apr;100(4):483-90. doi: 10.7326/0003-4819-100-4-483. PMID 6703540
- [Result] Trager K, Radermacher P. Catecholamines in the treatment of septic shock: effects beyond perfusion. Crit Care Resusc. 2003 Dec;5(4):270-6. PMID 16563117
- [Result] Hartmann C, Radermacher P, Wepler M, Nussbaum B. Non-Hemodynamic Effects of Catecholamines. Shock. 2017 Oct;48(4):390-400. doi: 10.1097/SHK.0000000000000879. PMID 28915214
- [Result] Hou T, Zhang R, Jian C, Ding W, Wang Y, Ling S, Ma Q, Hu X, Cheng H, Wang X. NDUFAB1 confers cardio-protection by enhancing mitochondrial bioenergetics through coordination of respiratory complex and supercomplex assembly. Cell Res. 2019 Sep;29(9):754-766. doi: 10.1038/s41422-019-0208-x. Epub 2019 Jul 31. PMID 31366990
- [Result] Banks L, Wells GD, McCrindle BW. Cardiac energy metabolism is positively associated with skeletal muscle energy metabolism in physically active adolescents and young adults. Appl Physiol Nutr Metab. 2014 Mar;39(3):363-8. doi: 10.1139/apnm-2013-0312. Epub 2013 Oct 9. PMID 24552379
- [Result] Gertz EW, Wisneski JA, Stanley WC, Neese RA. Myocardial substrate utilization during exercise in humans. Dual carbon-labeled carbohydrate isotope experiments. J Clin Invest. 1988 Dec;82(6):2017-25. doi: 10.1172/JCI113822. PMID 3198763
- [Result] Vieillard-Baron A, Caille V, Charron C, Belliard G, Page B, Jardin F. Actual incidence of global left ventricular hypokinesia in adult septic shock. Crit Care Med. 2008 Jun;36(6):1701-6. doi: 10.1097/CCM.0b013e318174db05. PMID 18496368
- [Result] Bouhemad B, Nicolas-Robin A, Arbelot C, Arthaud M, Feger F, Rouby JJ. Isolated and reversible impairment of ventricular relaxation in patients with septic shock. Crit Care Med. 2008 Mar;36(3):766-74. doi: 10.1097/CCM.0B013E31816596BC. PMID 18431265
- [Result] Bouhemad B, Nicolas-Robin A, Arbelot C, Arthaud M, Feger F, Rouby JJ. Acute left ventricular dilatation and shock-induced myocardial dysfunction. Crit Care Med. 2009 Feb;37(2):441-7. doi: 10.1097/CCM.0b013e318194ac44. PMID 19114917
- [Result] Kumar A, Bunnell E, Lynn M, Anel R, Habet K, Neumann A, Parrillo JE. Experimental human endotoxemia is associated with depression of load-independent contractility indices: prevention by the lipid a analogue E5531. Chest. 2004 Sep;126(3):860-7. doi: 10.1378/chest.126.3.860. PMID 15364767
- [Result] Vincent JL, Gris P, Coffernils M, Leon M, Pinsky M, Reuse C, Kahn RJ. Myocardial depression characterizes the fatal course of septic shock. Surgery. 1992 Jun;111(6):660-7. PMID 1595062
- [Result] Turner A, Tsamitros M, Bellomo R. Myocardial cell injury in septic shock. Crit Care Med. 1999 Sep;27(9):1775-80. doi: 10.1097/00003246-199909000-00012. PMID 10507597
- [Result] Chagnon F, Metz CN, Bucala R, Lesur O. Endotoxin-induced myocardial dysfunction: effects of macrophage migration inhibitory factor neutralization. Circ Res. 2005 May 27;96(10):1095-102. doi: 10.1161/01.RES.0000168327.22888.4d. Epub 2005 May 5. PMID 15879312
- [Result] Parrillo JE, Burch C, Shelhamer JH, Parker MM, Natanson C, Schuette W. A circulating myocardial depressant substance in humans with septic shock. Septic shock patients with a reduced ejection fraction have a circulating factor that depresses in vitro myocardial cell performance. J Clin Invest. 1985 Oct;76(4):1539-53. doi: 10.1172/JCI112135. PMID 4056039
- [Result] Duncan DJ, Yang Z, Hopkins PM, Steele DS, Harrison SM. TNF-alpha and IL-1beta increase Ca2+ leak from the sarcoplasmic reticulum and susceptibility to arrhythmia in rat ventricular myocytes. Cell Calcium. 2010 Apr;47(4):378-86. doi: 10.1016/j.ceca.2010.02.002. Epub 2010 Mar 12. PMID 20227109
- [Result] Wu AH. Increased troponin in patients with sepsis and septic shock: myocardial necrosis or reversible myocardial depression? Intensive Care Med. 2001 Jun;27(6):959-61. doi: 10.1007/s001340100970. No abstract available. PMID 11497152
- [Result] Tavernier B, Li JM, El-Omar MM, Lanone S, Yang ZK, Trayer IP, Mebazaa A, Shah AM. Cardiac contractile impairment associated with increased phosphorylation of troponin I in endotoxemic rats. FASEB J. 2001 Feb;15(2):294-6. doi: 10.1096/fj.00-0433fje. Epub 2000 Dec 8. PMID 11156941
- [Result] Kakihana Y, Ito T, Nakahara M, Yamaguchi K, Yasuda T. Sepsis-induced myocardial dysfunction: pathophysiology and management. J Intensive Care. 2016 Mar 23;4:22. doi: 10.1186/s40560-016-0148-1. eCollection 2016. PMID 27011791
- [Result] Murashige D, Jang C, Neinast M, Edwards JJ, Cowan A, Hyman MC, Rabinowitz JD, Frankel DS, Arany Z. Comprehensive quantification of fuel use by the failing and nonfailing human heart. Science. 2020 Oct 16;370(6514):364-368. doi: 10.1126/science.abc8861. PMID 33060364
- [Result] Dhainaut JF, Huyghebaert MF, Monsallier JF, Lefevre G, Dall'Ava-Santucci J, Brunet F, Villemant D, Carli A, Raichvarg D. Coronary hemodynamics and myocardial metabolism of lactate, free fatty acids, glucose, and ketones in patients with septic shock. Circulation. 1987 Mar;75(3):533-41. doi: 10.1161/01.cir.75.3.533. PMID 3815765
- [Result] Tessier JP, Thurner B, Jungling E, Luckhoff A, Fischer Y. Impairment of glucose metabolism in hearts from rats treated with endotoxin. Cardiovasc Res. 2003 Oct 15;60(1):119-30. doi: 10.1016/s0008-6363(03)00320-1. PMID 14522413
- [Result] Kreymann G, Grosser S, Buggisch P, Gottschall C, Matthaei S, Greten H. Oxygen consumption and resting metabolic rate in sepsis, sepsis syndrome, and septic shock. Crit Care Med. 1993 Jul;21(7):1012-9. doi: 10.1097/00003246-199307000-00015. PMID 8319458
- [Result] Panitchote A, Thiangpak N, Hongsprabhas P, Hurst C. Energy expenditure in severe sepsis or septic shock in a Thai Medical Intensive Care Unit. Asia Pac J Clin Nutr. 2017;26(5):794-797. doi: 10.6133/apjcn.072016.10. PMID 28802287
- [Result] Chagnon F, Bentourkia M, Lecomte R, Lessard M, Lesur O. Endotoxin-induced heart dysfunction in rats: assessment of myocardial perfusion and permeability and the role of fluid resuscitation. Crit Care Med. 2006 Jan;34(1):127-33. doi: 10.1097/01.ccm.0000190622.02222.df. PMID 16374166
- [Result] Levy RJ, Piel DA, Acton PD, Zhou R, Ferrari VA, Karp JS, Deutschman CS. Evidence of myocardial hibernation in the septic heart. Crit Care Med. 2005 Dec;33(12):2752-6. doi: 10.1097/01.ccm.0000189943.60945.77. PMID 16352955
- [Result] Szokodi I, Tavi P, Foldes G, Voutilainen-Myllyla S, Ilves M, Tokola H, Pikkarainen S, Piuhola J, Rysa J, Toth M, Ruskoaho H. Apelin, the novel endogenous ligand of the orphan receptor APJ, regulates cardiac contractility. Circ Res. 2002 Sep 6;91(5):434-40. doi: 10.1161/01.res.0000033522.37861.69. PMID 12215493
- [Result] Berry MF, Pirolli TJ, Jayasankar V, Burdick J, Morine KJ, Gardner TJ, Woo YJ. Apelin has in vivo inotropic effects on normal and failing hearts. Circulation. 2004 Sep 14;110(11 Suppl 1):II187-93. doi: 10.1161/01.CIR.0000138382.57325.5c. PMID 15364861
- [Result] Farkasfalvi K, Stagg MA, Coppen SR, Siedlecka U, Lee J, Soppa GK, Marczin N, Szokodi I, Yacoub MH, Terracciano CM. Direct effects of apelin on cardiomyocyte contractility and electrophysiology. Biochem Biophys Res Commun. 2007 Jun 15;357(4):889-95. doi: 10.1016/j.bbrc.2007.04.017. Epub 2007 Apr 12. PMID 17466269
- [Result] Chamberland C, Barajas-Martinez H, Haufe V, Fecteau MH, Delabre JF, Burashnikov A, Antzelevitch C, Lesur O, Chraibi A, Sarret P, Dumaine R. Modulation of canine cardiac sodium current by Apelin. J Mol Cell Cardiol. 2010 Apr;48(4):694-701. doi: 10.1016/j.yjmcc.2009.12.011. Epub 2009 Dec 28. PMID 20036246
- [Result] Li Z, He Q, Wu C, Chen L, Bi F, Zhou Y, Shan H. Apelin shorten QT interval by inhibiting Kir2.1/IK1 via a PI3K way in acute myocardial infarction. Biochem Biophys Res Commun. 2019 Sep 17;517(2):272-277. doi: 10.1016/j.bbrc.2019.07.041. Epub 2019 Jul 23. PMID 31349969
- [Result] Alfarano C, Foussal C, Lairez O, Calise D, Attane C, Anesia R, Daviaud D, Wanecq E, Parini A, Valet P, Kunduzova O. Transition from metabolic adaptation to maladaptation of the heart in obesity: role of apelin. Int J Obes (Lond). 2015 Feb;39(2):312-20. doi: 10.1038/ijo.2014.122. Epub 2014 Jul 16. PMID 25027224
- [Result] Mehrotra D, Wu J, Papangeli I, Chun HJ. Endothelium as a gatekeeper of fatty acid transport. Trends Endocrinol Metab. 2014 Feb;25(2):99-106. doi: 10.1016/j.tem.2013.11.001. Epub 2013 Dec 3. PMID 24315207
- [Result] Feng J, Zhao H, Du M, Wu X. The effect of apelin-13 on pancreatic islet beta cell mass and myocardial fatty acid and glucose metabolism of experimental type 2 diabetic rats. Peptides. 2019 Apr;114:1-7. doi: 10.1016/j.peptides.2019.03.006. Epub 2019 Apr 4. PMID 30954534
- [Result] Saleme B, Das SK, Zhang Y, Boukouris AE, Lorenzana Carrillo MA, Jovel J, Wagg CS, Lopaschuk GD, Michelakis ED, Sutendra G. p53-Mediated Repression of the PGC1A (PPARG Coactivator 1alpha) and APLNR (Apelin Receptor) Signaling Pathways Limits Fatty Acid Oxidation Energetics: Implications for Cardio-oncology. J Am Heart Assoc. 2020 Aug 4;9(15):e017247. doi: 10.1161/JAHA.120.017247. Epub 2020 Jul 29. No abstract available. PMID 32750288
- [Result] Rudiger A, Dyson A, Felsmann K, Carre JE, Taylor V, Hughes S, Clatworthy I, Protti A, Pellerin D, Lemm J, Claus RA, Bauer M, Singer M. Early functional and transcriptomic changes in the myocardium predict outcome in a long-term rat model of sepsis. Clin Sci (Lond). 2013 Mar;124(6):391-401. doi: 10.1042/CS20120334. PMID 22988837
- [Result] Chagnon F, Coquerel D, Salvail D, Marsault E, Dumaine R, Auger-Messier M, Sarret P, Lesur O. Apelin Compared With Dobutamine Exerts Cardioprotection and Extends Survival in a Rat Model of Endotoxin-Induced Myocardial Dysfunction. Crit Care Med. 2017 Apr;45(4):e391-e398. doi: 10.1097/CCM.0000000000002097. PMID 27571457
- [Result] Coquerel D, Chagnon F, Sainsily X, Dumont L, Murza A, Cote J, Dumaine R, Sarret P, Marsault E, Salvail D, Auger-Messier M, Lesur O. ELABELA Improves Cardio-Renal Outcome in Fatal Experimental Septic Shock. Crit Care Med. 2017 Nov;45(11):e1139-e1148. doi: 10.1097/CCM.0000000000002639. PMID 28777197
- [Result] Frier BC, Williams DB, Wright DC. The effects of apelin treatment on skeletal muscle mitochondrial content. Am J Physiol Regul Integr Comp Physiol. 2009 Dec;297(6):R1761-8. doi: 10.1152/ajpregu.00422.2009. Epub 2009 Sep 30. PMID 19793954
- [Result] Masse MH, Richard MA, D'Aragon F, St-Arnaud C, Mayette M, Adhikari NKJ, Fraser W, Carpentier A, Palanchuck S, Gauthier D, Lanthier L, Touchette M, Lamontagne A, Chenard J, Mehta S, Sansoucy Y, Croteau E, Lepage M, Lamontagne F. Early Evidence of Sepsis-Associated Hyperperfusion-A Study of Cerebral Blood Flow Measured With MRI Arterial Spin Labeling in Critically Ill Septic Patients and Control Subjects. Crit Care Med. 2018 Jul;46(7):e663-e669. doi: 10.1097/CCM.0000000000003147. PMID 29629988